CLINICAL TRIAL: NCT04795778
Title: The Validity and Reliability of FIT-HaNSA (Functional Impairment Test-Hand and Neck/Shoulder/Arm) in Breast Cancer Patients
Brief Title: The Validity and Reliability of FIT-HaNSA in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Principal Investigator, Gazi University
Other Study IDs: IAyas2
Record Dates: First submitted 2021-03-11; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; FIT-HaNSA; Upper Extremity Dysfunction
Keywords: Breast Cancer; FIT-HaNSA; Upper Extremity Dysfunction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with breast cancer: Breast cancer patients with or without breast cancer surgery, with or without mastectomy, with or without lymphedema
- Control group: Healty individuals with no disease

SUMMARY:
Breast cancer is the most common type of cancer among women and covers 25% of all cancers. After mastectomy and reconstruction, many patients develop various upper extremity complications such as joint movement limitation, pain, lymphedema, and axillary cord. Because of such upper extremity problems, evaluation and treatment of upper extremity functions are important. Upper extremity functions are generally evaluated with questionnaires filled out by the patients themselves and which reflect their own perspectives subjectively. However, these questionnaires cannot reflect the observations and evaluations of the clinicians. Performance tests are important for clinicians to make decisions.

With this study, we want to examine the usability of the FIT-HaNSA test in the evaluation of upper extremity functions in patients with breast cancer. Our hypothesis; The FıtHaNSA test is successful in evaluating the upper extremity function in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Those whose treatments for breast cancer have been completed 18 years and over

Exclusion Criteria:

* Have a history of upper extremity surgery, excluding breast cancer surgery Have a history of upper extremity trauma Those who have orthopedic, neurological, rheumatological or cognitive impairments that may interfere with the application of the test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients referred to physiotherapy and rehabilitation from Gazi University hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
FIT-HaNSA test for upper extremity performance | For the patient group; at least 3 months after all treatments have been completed
  FIT-HaNSA protocol includes 3 steps.In the first step of the test 3 weights of 1kg are placed on the shelf at the waist level of the individual at 10 cm intervals.The person moves these weights in rows to the 25 cm upper rack and then place them back on the lower rack.The person is asked to continue this process for 5 minutes.In the second step of the test, the first shelf is placed at eye level, the second shelf is placed 25 cm below it and the procedures in the first step are repeated.In the 3rd step, a wooden plate with 3 holes is placed perpendicular to the shelf at eye level of the individual.The hole in the middle is left empty by placing nuts and bolts in the first and third holes before. The individual must return to the starting point in order by attaching the bolt in the first hole to the second hole, the bolt in the third hole to the first hole and finally the bolt in the second hole to the third hole and this process is 5 minutes.
Upper extremity disability | For the patient group; at least 3 months after all treatments have been completed
  Upper extremity disability will be evaluated with DASH questionnaire (Disabilities of the Arm, Shoulder and Hand). It is a questionnaire consisting of 30 questions that evaluates the dysfunctions of the entire upper extremity. It consists of questions evaluating the degree of difficulty in performing different activities using the upper extremity in daily life (21 questions), pain, numbness, joint stiffness and weakness symptoms (5 questions), social life, sleep, work and psychological status (4 questions) in the last week.
Upper extremity functionality | For the patient group; at least 3 months after all treatments have been completed
  Upper extremity functionality will be evaluated with Upper Extremity Functional Index (UEFI). It is a questionnaire consisting of 20 questions that questions the functional difficulty of the upper extremity in daily life activities. Each question is scored between 0 and 4 (0: extremely difficult, 4: no difficulty).
Shoulder disability | For the patient group; at least 3 months after all treatments have been completed
  Shoulder disability will be evaluated with Shoulder Pain and Disabilty Index (SPADI). The scale, which consists of 13 questions in total, has two subsections as pain and disability. The pain section consists of 5 questions describing the pain of the patient, and the disability section consists of 8 questions that indicate the degree of difficulty experienced when using the upper extremity. Each question is scored from 0 to 10 (0 is no difficulty, 10 is very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: inci ayas, Study Director — Gazi University
Locations (1):
- Inci Ayas, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only study officials will be able to view patient data The statistical analysis will also be done by the study officials.